CLINICAL TRIAL: NCT04658121
Title: SARS-CoV-2 Prevalence Study
Brief Title: SARS-CoV-2/COVID-19 Prevalence Study
Status: Completed | Type: Observational
Sponsor: COVID-19 Prevention Network (Network)
Responsible Party: Sponsor
Other Study IDs: CoVPN 5002
Record Dates: First submitted 2020-11-19; First posted 2020-12-08 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood collection, nasal mid-turbinate swab, and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Senior Living Facilities: Adults residing in senior living facilities (nursing homes, assisted or independent living facilities)
- Outpatient Healthcare Facilities: Adults attending outpatient healthcare in neighborhoods of selected research sites
- General Communities: Adults and children (>2 months of age) in neighborhoods of selected research sites

SUMMARY:
The COVID-19 Prevention Network (CoVPN) is doing a study to estimate the number of people who have or have had the SARS-CoV-2 virus in different communities in the United States. This study is being done to help determine the best places to perform future research studies that will test new drugs for treatment or prevention of COVID-19.

DETAILED DESCRIPTION:
Design:

Cross-sectional surveys of (1) adults residing in senior living facilities and attending outpatient healthcare facilities, and (2) the general population in each selected research site community.

Population:

1. Adults residing in senior living facilities (nursing homes, assisted or independent living facilities) and attending outpatient healthcare facilities in neighborhoods of selected research sites
2. Adults and children (> 2 months of age) in neighborhoods of selected research sites

Study Size:

For each research site, up to 3,920 individuals will be enrolled from one, two, or all three of the following populations (must include at least community venues):

1. senior living facilities (nursing homes, assisted or independent living facilities; n = 500)
2. outpatient healthcare facilities (n = 500)
3. community venues distributed across four age categories (0-17, 18-39, 40-59, 60+ years) (n = 730 per stratum or 2920)

Total sample size = 3,920 x up to 20 clinical research sites

Study Duration:

Approximately sixteen (16) months for overall project. Two (2) months for protocol development and institutional review board (IRB) approval, followed by:

1. Facility-based surveys: 12 months (3 months for site preparation and initiation, 3 months for enrollment/sample collection, 4 months for shipping and laboratory testing*, 2 months for close-out), concurrent with
2. Time-location sampling (TLS) surveys: 14 months (3 months for site preparation and initiation, 6 months for enrollment/sample collection, 6 months for shipping and laboratory testing*, 2 months for close-out)

   * Some activities will be concurrent with enrollment

Study Location:

Catchment areas surrounding US-based Clinical Research Sites (CRSs) of the: HIV Prevention Trials Network (HPTN), HIV Vaccine Trials Network (HVTN), Infectious Diseases Clinical Research Consortium (IDCRC), International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT), and the AIDS Clinical Trials Group (ACTG); to be specified in the Site Announcement Memo

Study Methods:

Blood collection for SARS-CoV-2 antibody testing and characterization of the serologic response to SARS-CoV-2 infection; nasal mid-turbinate swab collection for SARS-CoV-2 RNA testing; collection of saliva in a subset of participants to evaluate the performance of diagnostic SARS-CoV-2 assays using these matrices; administration of tablet-based survey. Medical records abstraction for senior living facility participants who are unable to respond to the study survey.

ELIGIBILITY:
Inclusion Criteria:

Adults residing in senior living facilities or attending outpatient healthcare facilities:

* At least 18 years of age
* Willing and able to provide informed consent or consent has been provided by legal representative (for those with mental incapacity in senior living facilities)
* Recruited from a selected facility

Adults and children from select neighborhoods of research site communities:

* Adults and children > 2 months of age
* For individuals < 18 years old, a guardian must be present (in person or by phone for those 15 - 17 years old)
* Willing and able to provide consent (or assent for individuals 7-17 years old, parent/guardian will provide consent for all minors)
* Recruited from a selected venue

Exclusion Criteria:

* Previous enrollment in this study, either from the same or another CRS community.
* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults residing in nursing homes or attending outpatient healthcare facilities in neighborhoods of selected research sites. Adults and children (>2 month of age) in neighborhoods of selected research sites.
Sampling Method: Probability Sample
Enrollment: 26741 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of SARS-CoV-2 IgG seropositivity among individuals in communities surrounding selected NIAID clinical research sites | Baseline

SECONDARY OUTCOMES:
To estimate prevalence of SARS-CoV-2 infection based on results of SARS-CoV-2 RNA testing | Baseline
To estimate prevalence of SARS-CoV-2 infection by presence versus absence of symptoms consistent with COVID-19 | Baseline
To estimate seroprevalence of SARS-CoV-2 | Baseline
  Among:
  1. Those without past or current symptoms consistent with COVID-19
  2. Those with no prior positive SARS-CoV-2 testing, but who report close contact with confirmed or presumed cases
  3. Those with history of co-morbid medical conditions
To assess association between demographic, clinical and social factors with SARS-CoV-2 infection and seroprevalence, with particular interest in racial and ethnic health disparities. | Baseline
  Logistic regression using survey weights will be used to infer associations between the hypothesized socioeconomic, demographic and clinical predictors of SARS-CoV-2 infection and seroprevalence.
To estimate potential size of populations for referral to COVID-19 prevention and treatment studies | Baseline
To assess knowledge, attitudes, and behavior about SARS-CoV-2 and COVID-19 through a study questionnaire | Baseline
To assess performance characteristics of PCR-based and serologic SARS-CoV-2 tests using saliva samples | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justman, MD, Study Chair — Departments of Epidemiology and Medicine, Columbia University
Locations (15):
- United States (14):
  - Children's Hospital Colorado CRS, Aurora, Colorado
  - U of Miami, IDRU at Jackson Memorial Hospital CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - UIC Project Wish CRS, Chicago, Illinois
  - New Orleans Adolescent Trials Unit CRS, New Orleans, Louisiana
  - John's Hopkins CRS, Baltimore, Maryland
  - New Jersey Medical School CRS, Newark, New Jersey
  - Harlem Prevention, New York, New York
  - Physicians & Surgeons CRS, New York, New York
  - Bronx Prevention Center, New York, New York
  - Cincinnati CRS, Cincinnati, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- St. Louis University VTEU-CAIMED-PHSU, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: COVID-19 Nursing Home Data [Internet].2020 [cited 06/08/2020] — http://data.cms.gov/stories/s/COVID-19-Nursing-Home-Data/bkwz-xpvg

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04658121/Prot_ICF_000.pdf